CLINICAL TRIAL: NCT00001598
Title: Dehydroepiandrosterone (DHEA) Treatment for Sjogren's Syndrome
Brief Title: DHEA Treatment for Sjogren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970123; 97-D-0123
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-06

CONDITIONS: Lacrimal Apparatus Disease; Salivary Gland Disease; Sjogren's Syndrome; Xerostomia
Keywords: Xerostomia; Autoimmunity; Salivary Glands; Androgen Therapy; Lacrimal Function; DHEA; Sjogren's Syndrome; Dehydroepiandrosterone
MeSH Terms: conditions — Lacrimal Apparatus Diseases; Salivary Gland Diseases; Sjogren's Syndrome; Xerostomia; Autoimmune Diseases | interventions — Dehydroepiandrosterone

INTERVENTIONS:
Drug: Dehydroepiandrosterone

SUMMARY:
This study will evaluate the effectiveness of the male hormone dehydroepiandrosterone (DHEA) in treating Sjogren's syndrome. This autoimmune disorder, in which the immune system attacks the salivary glands and tear glands, affects primarily women. Patients' eyes and mouth become drier over time, and can lead to problems such as serious tooth decay and eye irritations. Sex hormones seem to influence the immune response and may help decrease disease severity. DHEA has benefited some patients with two other autoimmune diseases, rheumatoid arthritis and systemic lupus erythematosus.

Women 18 to 75 years of age with Sjogren's syndrome may be eligible for this 7-month study. At the initial visit, candidates will have a physical examination, routine blood and urine tests and eye and dental examinations, including a test to measure saliva production for screening purposes and to establish baseline values for participants.

Those enrolled in the study will be randomly assigned to take either DHEA or placebo (look-alike tablet with no active ingredient) once a day for 6 months and will be monitored with follow-up visits at months 1, 3, 6 and 7. Physical examination, blood tests and urinalysis will be repeated at months 1, 3, 6 and 7; saliva will be collected at months 3, 6 and 7; and eyes will be examined at 3 and 6 months. Because hormone changes may have both physical and emotional effects, patients will be asked questions about their mood, symptoms and side effects of treatment.

It is not known if Sjogren's syndrome is associated with osteoporosis (bone thinning), but since this condition occurs in other autoimmune disorders, patient's bone density will be measured at the first visit, and blood drawn at 3 and 6 months will be tested for various substances associated with changes in bone density. A 24-hour urine collection at the first visit and later urine tests will also be tested for substances associated with bone thinning.

DETAILED DESCRIPTION:
Primary Sjogren's syndrome (SS) is an autoimmune disease chiefly affecting the exocrine glands. One of the most troublesome manifestations of SS is severe salivary gland dysfunction. There is no accepted treatment for the underlying autoimmune reactivity or the salivary gland dysfunction in SS. SS, as well as many other autoimmune diseases, predominantly affects women. Although sex hormones do not cause SS or other autoimmune disease, they appear to influence immunological responses and ultimately the severity of disease. We propose to test the effects of dehydroepiandrosterone (DHEA), a mildly androgenic adrenal hormone, on lacrimal and salivary gland function in SS. In a randomized, double-masked, outpatient protocol, patients will receive DHEA for 6 months. Efficacy of treatment will be assessed by monitoring salivary and lacrimal function, serological markers of autoimmune activity, and subjective reports of local and systemic symptoms.

ELIGIBILITY:
Females with a diagnosis of Primary Sjogren's Syndrome.

No history of breast cancer.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28
Dates: Start 1997-05; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Johnson JT, Ferretti GA, Nethery WJ, Valdez IH, Fox PC, Ng D, Muscoplat CC, Gallagher SC. Oral pilocarpine for post-irradiation xerostomia in patients with head and neck cancer. N Engl J Med. 1993 Aug 5;329(6):390-5. doi: 10.1056/NEJM199308053290603. PMID 8326972
- [Background] van Vollenhoven RF, Engleman EG, McGuire JL. An open study of dehydroepiandrosterone in systemic lupus erythematosus. Arthritis Rheum. 1994 Sep;37(9):1305-10. doi: 10.1002/art.1780370906. PMID 7945493
- [Background] Lucas JA, Ahmed SA, Casey ML, MacDonald PC. Prevention of autoantibody formation and prolonged survival in New Zealand black/New Zealand white F1 mice fed dehydroisoandrosterone. J Clin Invest. 1985 Jun;75(6):2091-3. doi: 10.1172/JCI111929. PMID 3159756